CLINICAL TRIAL: NCT05153408
Title: A Phase 1/2 Study of the Highly Selective EGFR Inhibitor, BLU-701, in Patients With EGFR-Mutant Non-Small Cell Lung Cancer
Brief Title: (HARMONY) Study of BLU-701 in EGFR-mutant NSCLC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Blueprint Medicines Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BLU-701-1101
Record Dates: First submitted 2021-11-30; First posted 2021-12-10 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Lung Neoplasm; Carcinoma, Non-Small-Cell Lung; Respiratory Tract Neoplasms; Neoplasms; Neoplasms by Site; Lung Diseases; Respiratory Tract Diseases; Carcinoma, Bronchogenic; Bronchial Neoplasms; Adenocarcinoma; Carcinoma; Neoplasms by Histologic Type; Neoplasms, Nerve Tissue; EGFR C797S; EGFR C797A; EGFR L858R; EGFR Exon 19 Deletion; EGFR Gene Mutation; EGF-R Positive Non-Small Cell Lung Cancer; EGFR Mutation Resulting in Tyrosine Kinase Inhibitor Resistance; EGFR Activating Mutation; Thoracic Neoplasms; Antineoplastic Agents; Protein Kinase Inhibitors; EGFR C797G; EGFR C797X; Non Small Cell Lung Cancer
Keywords: Targeted therapy; EGFR; NSCLC; non-small cell lung cancer; EGFR mutant NSCLC
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Respiratory Tract Neoplasms; Neoplasms; Neoplasms by Site; Lung Diseases; Respiratory Tract Diseases; Carcinoma, Bronchogenic; Bronchial Neoplasms; Adenocarcinoma; Carcinoma; Neoplasms by Histologic Type; Neoplasms, Nerve Tissue; Thoracic Neoplasms | interventions — osimertinib; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1A: BLU-701 as monotherapy (Experimental): Phase 1 dose escalation of BLU-701 as monotherapy at various dose levels
  Interventions: Drug: BLU-701
- Part 1B: BLU-701 with osimertinib (Experimental): BLU-701 in combination with osimertinib 40 mg or 80 mg tablets for oral administration
  Interventions: Drug: BLU-701; Drug: osimertinib
- Part 1C: BLU-701 with platinum-based chemotherapy (Experimental): BLU-701 in combination with platinum-based chemotherapy (carboplatin and pemetrexed):
  Carboplatin - IV infusion dosed to target AUC of 5-6 mg/mL min q3w
  Pemetrexed - IV infusion dosed to 500 mg/m2 q3w
  Interventions: Drug: BLU-701; Drug: carboplatin; Drug: pemetrexed
- Part 2A: BLU-701 as monotherapy (Experimental): Phase 2 expansion group for BLU-701 as monotherapy at a dose determined during Part 1A in patients harboring the EGFR C797X resistance mutation
  Interventions: Drug: BLU-701

INTERVENTIONS:
Drug: BLU-701 — BLU-701 for oral administration
Drug: osimertinib — Osimertinib tablets for oral administration
  Other Names: Tagrisso
  Arms: Part 1B: BLU-701 with osimertinib
Drug: carboplatin — IV infusion of carboplatin
  Arms: Part 1C: BLU-701 with platinum-based chemotherapy
Drug: pemetrexed — IV infusion of pemetrexed
  Arms: Part 1C: BLU-701 with platinum-based chemotherapy

SUMMARY:
This is a Phase 1/2, open-label, first-in-human (FIH) study is designed to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and antitumor activity of BLU-701 as monotherapy or in combination with either osimertinib or platinum-based chemotherapy in patients with EGFRm NSCLC.

DETAILED DESCRIPTION:
The study was planned to include an initial Phase 1 portion to determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of BLU-701 as monotherapy (Part 1A; initially in a once daily (QD) regimen with the option to evaluate twice daily (BID) dosing if supported by emerging PK and safety data), as well as additional dose-escalation portions to determine the RP2D of BLU-701 in combination with osimertinib (Part 1B) or in combination with carboplatin and pemetrexed (Part 1C). A Phase 2 part was planned to further evaluate the efficacy and safety of BLU-701 as monotherapy at RP2D (Part 2A). Phase 1 Part 1 A was initiated; however, the study was terminated prior to establishing BLU-701 MTD and/or RP2D.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age at the time of signing the informed consent.
2. Pathologically confirmed metastatic NSCLC.
3. Tumor mutation profile determined locally via next generation sequencing (NGS), using tumor tissue (preferably from a progressing lesion) and/or ctDNA in plasma. For Phase 1, it is preferable that samples used for analysis be obtained during or after disease progression on the last EGFR-targeted TKI received. For Phase 2, samples used for analysis must be obtained during or after disease progression on the last EGFR-targeted TKI received.

   1. All Parts: activating EGFR mutation (Ex19Del or L858R)
   2. Part 2A: Tumor must additionally harbor an EGFR C797X resistance mutation.
4. Previously received:

   1. Part 1A and 2A: At least 1 prior third-generation EGFR-targeted TKI, such as osimertinib
   2. Part 1B: Patients must have experienced progressive disease while on osimertinib, were able to tolerate prior osimertinib 80 mg QD dose, and continuing on osimertinib is deemed to be in the patient's best interests in the opinion of the Investigator.

      Patients who have discontinued osimertinib may be eligible, if no more than 6 weeks elapse between the discontinuation of prior osimertinib and resumption of osimertinib on study.
   3. Part 1C: At least 1 prior EGFR-targeted TKI
5. Willing to provide pretreatment tumor sample (either an archival sample or a sample obtained by pretreatment biopsy. For Phase 1, it is preferable that pretreatment tumor sample be obtained from a progressing lesion and during or after disease progression on the last EGFR-targeted TKI received. For Phase 2, pretreatment tumor sample must be obtained during or after disease progression on the last EGFR-targeted TKI treatment received. Patients without appropriate archival tissue available, where biopsy is not considered safe and/or medically feasible, may be discussed with the study medical monitor and approved for enrollment on a case-by-case basis.
6. Part 2A: at least 1 measurable target lesion per RECIST 1.1 as assessed by the Investigator
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
8. Agrees to use contraception consistent with local regulations

Exclusion Criteria:

1. Have disease that is suitable for local therapy administered with curative intent.
2. Have tumor that harbors EGFR T790M mutation or any additional known driver alterations (including but not limited to, EGFR exon 20 insertions, or pathologic abnormalities of KRAS, BRAF V600E, NTRK1/2/3, HER2, ALK, ROS1, MET, or RET).
3. Have NSCLC with mixed cell histology or a tumor with known histologic transformation (NSCLC to SCLC, SCLC to NSCLC, or epithelial to mesenchymal transition).
4. Have received the following anticancer therapy:

   1. Any third-generation EGFR TKI (such as osimertinib) within 7 days prior to the planned first dose of study drug. Note: patients in Part 1B do not require a wash-out period for osimertinib.
   2. Part 2A: Previous therapy with first- or second-generation EGFR TKI, such as erlotinib, gefitinib, afatinib or dacomitinib.
   3. Part 1C: Prior platinum-based chemotherapy for advanced or metastatic disease.
   4. Any immunotherapy or other antibody therapy (including EGFR-targeted antibodies or bi-specific antibodies) within 21 days prior to the first dose of study drug.
   5. Any other systemic anticancer therapy within 14 days or 5 half-lives prior to the first dose of study drug, whichever is the shortest, but with a minimum of 7 days in all circumstances. BLU-701 may be started within these washout periods if considered by the Investigator to be safe and within the best interest of the patient, with prior Sponsor approval.
5. Radiotherapy to a large field or including a vital organ (including whole brain radiotherapy or stereotactic radiosurgery to brain) within 14 days before the first dose of study drug. Radiotherapy to a focal site of disease that did not include a vital organ (such as a limb) within 7 days before the first dose of study drug.
6. Have CNS metastases or spinal cord compression that is associated with progressive neurological symptoms or requires increasing doses of corticosteroids to control the CNS disease. If a patient requires corticosteroids for management of CNS disease, the dose must have been stable for the 2 weeks preceding treatment. Asymptomatic CNS and leptomeningeal disease is allowed and, when measurable, should be captured as target lesions.
7. Have any of the following laboratory abnormalities on last laboratory assessment prior to initiation of study drug (i.e., C1D1 or Screening):

   1. Absolute neutrophil count (ANC) <1.0×109/L (for patients in Part 1C: <1.5×109/L)
   2. Platelet count <75×109/L (for patients in Part 1C: <100×109/L)
   3. Hemoglobin ≤8.0 g/dL (red blood cell transfusion and erythropoietin may be used to reach at least 8.0 g/dL but must have been administered at least 2 weeks prior to the first dose of study drug).
   4. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2.5× the upper limit of normal (ULN) if no hepatic metastases are present; >5× ULN if hepatic metastases are present.
   5. Total bilirubin >1.5× ULN; >3× ULN in presence of Gilbert's disease.
   6. Estimated (Cockroft-Gault formula, Appendix 1) or measured creatinine clearance <60 mL/min.
   7. International normalized ratio (INR) >2.3 or prothrombin time (PT) >6 seconds above ULN or a patient-specific INR or PT abnormality that the treating investigator considers clinically relevant and/or increases the risk for hemorrhage in that individual patient.
8. Have known intracranial hemorrhage and/or bleeding diatheses.
9. Have clinically active ongoing interstitial lung disease (ILD) of any etiology, including drug-induced ILD, and radiation pneumonitis within 28 days prior to initiation of study treatment. Grade 1 asymptomatic ILD is not exclusionary.
10. Have any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 or that have not resolved to baseline at the time of starting the study. Exceptions include alopecia and fatigue, and, upon discussion with and approval by the Medical Monitor, other toxicities that are not thought to present a risk to patient safety.
11. Have mean resting QT interval corrected using Fridericia's formula (QTcF) >450 msec, a history of prolonged QT syndrome or Torsades de pointes, or a familial history of prolonged QT syndrome.
12. Have clinically significant, uncontrolled, cardiovascular disease including congestive heart failure Grade III or IV according to the New York Heart Association classification; myocardial infarction or unstable angina within the previous 6 months, uncontrolled hypertension, or clinically significant, uncontrolled arrhythmias, including bradyarrhythmia that may cause QT prolongation (e.g., Type II second degree heart block or third degree heart block).
13. Have history of another primary malignancy (other than completely resected carcinomas in situ) that has been diagnosed or required therapy within 2 years prior to initiation of study treatment. However, upon discussion with the Sponsor, patients who have another concurrent malignancy (not lung cancer) that is clinically stable and does not require tumor-directed treatment may be eligible to participate. Examples include, but are not limited to, completely resected basal cell carcinoma and squamous cell carcinoma of skin; curatively treated prostate cancer, breast cancer; and early gastric cancer cured by endoscopic mucosal resection or endoscopic submucosal dissection.
14. Have active, uncontrolled infection (viral, bacterial, or fungal), including tuberculosis, hepatitis B, hepatitis C, AIDS-related illness, or COVID19 infection. Controlled infections, including HIV and "cured" hepatitis C (no active fever, no evidence of systemic inflammatory response syndrome) that are stable on antiviral treatment are not exclusionary.
15. For Parts 1A, 1B, and 1C: have received neutrophil or platelet growth factor support within 14 days of the first dose of study drug.
16. Require treatment with a prohibited medication or herbal remedy that cannot be discontinued at least 2 weeks before the start of study drug administration. BLU-701 may be started within 14 days or 5 half-lives of these therapies if considered by the Investigator to be safe and within the best interest of the patient, with prior Sponsor approval.
17. Have major surgical procedure within 14 days of the first dose of study drug (procedures such as central venous catheter placement, tumor needle biopsy, and feeding tube placement are not considered major surgical procedures).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
[Phase 1] Determine the maximum tolerated dose (MTD) of BLU-701 monotherapy, BLU-701 in combination with osimertinib, and BLU-701 in combination with platinum-based chemotherapy | Up to 12 months
  MTD determination: dose limiting toxicity (DLT) rate
[Phase 1] Determine the recommended Phase 2 dose (RP2D) of BLU-701 monotherapy, BLU-701 in combination with osimertinib, and BLU-701 in combination with platinum-based chemotherapy | Up to 12 months
  RP2D determination: DLT, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary safety and antitumor activity data
[Phase 1] Overall safety profile | Up to 12 months
  Rate and severity of adverse events
[Phase 2] Overall response rate (ORR) | Up to 30 months
  ORR - the proportion of patients who experience a best response of confirmed CR or PR according to RECIST 1.1

SECONDARY OUTCOMES:
[Phase 1] Overall response rate (ORR) | Up to 12 months
  ORR - the proportion of patients who experience a best response of confirmed complete response (CR) or partial response (PR) according to RECIST 1.1
[Phase 1 and Phase 2] Duration of response (DOR) | Up to 42 months
  DOR - time from first documented response of CR or PR to the date of first documented progressive disease or death due to any cause, whichever occurs first
[Phase 1 and Phase 2] To characterize the PK profile of BLU-701 | Up to 42 months
  maximum plasma drug concentration (Cmax) time to maximum plasma drug concentration (Tmax) time of last quantifiable plasma drug concentration (Tlast) area under the plasma concentration versus time curve from time 0 to the end of the dosing interval (AUC0-24 for QD and AUC0-12 for BID) trough concentration (Ctrough) apparent volume of distribution (Vz/F) terminal elimination half-life (t½) apparent oral clearance(CL/F) accumulation ratio (R)
[Phase 1] To assess treatment-induced modulation of EGFR pathway biomarkers for BLU-701 monotherapy | Up to 42 months
  dual specificity phosphatase (DUSP6)
  sprouty RTK signaling antagonist 4 (SPRY4)
[Phase 2] Overall safety profile | Up to 42 months
  Rate and severity of adverse events
[Phase 2]Disease Control Rate (DCR) | Up to 42 months
  DCR - proportion of patients who experience a best response of CR, PR, or SD according to RECIST 1.1
[Phase 2] Clinical Benefit Rate (CBR) | Up to 42 months
  CBR - proportion of patients who experience a confirmed CR or PR, or SD with a duration of at least 16 weeks according to RECIST 1.1
[Phase 2] Progression Free Survival (PFS) | Up to 42 months
  PFS - time from the first dose of BLU-701 until the date of first documented PD or death due to any cause
[Phase 2] Overall Survival (OS) | Up to 42 months
  OS - time from the first dose of BLU-701 until the date of death due to any cause
[Phase 2] Central Nervous System Overall Response Rate (CNS-ORR) | Up to 42 months
  CNS-ORR - proportion of patients with measurable (target) intracranial metastases at baseline who experience a confirmed intracranial CR or PR according to RECIST 1.1 principles
[Phase 2] Central Nervous System Duration of Response (CNS-DOR) | Up to 42 months
  CNS-DOR - time from first documented intracranial CR or PR to the date of first documented intracranial PD
[Phase 2] Central Nervous System Progression Rate | Up to 42 months
  CNS progression rate - proportion of patients with CNS progression as a component of first disease progression on study
[Phase 2] To assess the effect of BLU-701 on cardiovascular intervals, including QT, and rhythm | Up to 42 months
  ECG parameters extracted from continuous 12-lead Holter recordings

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - New York University (NYU) Langone Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - NEXT Virginia, Fairfax, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No